CLINICAL TRIAL: NCT04131582
Title: Effect of a Quadruple Therapy on Pancreatic Islet Function, Insulin Resistance and Cardiovascular Function in Patients With Mixed Prediabetes and Obesity: Randomized Clinical Trial
Brief Title: Effect of Empagliflozin + Linagliptin + Metformin + Lifestyle in Patients With Prediabetes
Acronym: 4T
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Guanajuato (Other)
Collaborators: Hospital Regional de Alta Especialidad del Bajio (Other)
Responsible Party: Principal Investigator, Rodolfo Guardado Mendoza, Principal Investigator, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CI/HRAEB/2017/049
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Prediabetic State; Insulin Resistance
Keywords: prediabetes
MeSH Terms: conditions — Prediabetic State; Insulin Resistance | interventions — Linagliptin; Metformin; empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Assigned treatments will be delivered to the patients in identical envelopes by a person not involved in the trial; persons who evaluate the follow-up and outcomes will be masked to the treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin + linagliptin + metformin plus lifestyle (Experimental): Patients are randomized to receive for 12 months Linagliptin 2.5 mg + metformin 850 mg every 12 hours and empagliflozin 12.5 mg + metformin 850 mg every 12 hours. The start of the dose in this group will be gradual so that at the month of treatment the patient can be with the full doses. Together with this, patients will receive a lifestyle modification program seeking to reduce 5-7% of body weigh and increase physical activity to 90/150 min/week
  Interventions: Combination Product: Linagliptin + metformin and Empagliflozin + metformin
- Metformin plus lifestyle (Active Comparator): Patients are randomized to receive for 12 months Metformin 850 mg every 12 hours. The start of the dose in this group will be gradual so that at the month of treatment the patient can be with the complete dose. Together with this, patients will receive a lifestyle modification program seeking to reduce 5-7% of body weigh and increase physical activity to 90/150 min/week
  Interventions: Drug: Metformin

INTERVENTIONS:
Combination Product: Linagliptin + metformin and Empagliflozin + metformin — Linagliptin-Metformin 2.5/850mg once daily, Empagliflozin-Metformin 12.5/850mg one daily plus a lifestyle modification program based on nutritional assesment, physical activity prescription and general counseling
  Other Names: Trayenta Duo + Jardianz Duo
  Arms: Empagliflozin + linagliptin + metformin plus lifestyle
Drug: Metformin — Metformin 850mg twice daily plus a lifestyle modification program based on nutritional assesment, physical activity prescription and general counseling
  Arms: Metformin plus lifestyle

SUMMARY:
Type 2 diabetes is a worldwide epidemic disease, and preventive strategies are needed to face this health problem. The goal of this trial is to evaluate the effect of empagliflozin + linagliptin + metformin + lifestyle on physiopathological parameters, sush as glucose metabolism, insulin resistance, pancreatic beta cell function and cardiovascular function in patients with impaired fasting glucose plus impaired glucose tolerance, during 12 months

DETAILED DESCRIPTION:
The main goal of this clinical trial is to compare the effect of two different treatments during 12 months:

1. Lifestyle modification program + metformin 850 mg twice daily
2. Lifestyle modification program empagliflozin (12.5 mg) + metformin (850 mg) once daily plus linagliptin (2.5 mg) + metformin (850 mg) once daily On the following parameters, after 12 months of treatment

1) Glucose metabolism, evaluated by oral glucose tolerance test 2) Insulin resistance evaluated by the oral glucose tolerance 3) Insulin secretion, evaluated by the oral glucose tolerance 4) Pancreatic beta cell function, evaluated by the oral glucose tolerance test 5) Cardiovascular function, evaluated by standard echocardiography by left ventricular ejection fraction

All the patients will have a basal evaluation with an oral glucose tolerance test, lipid profile and body composition measurement by dual energy X-ray absorptiometry (DEXA). After the basal evaluation, if the patients results with impaired fasting glucose and impaired glucose tolerance, they will be invited to the intervention phase where they will be randomized to one of the two treatment groups.

Patients will have a follow-up visit every month to review the adherence to the lifestyle modification program and to the medication, and every 6 months an OGTT. After 12 months , patients will repeat the same evaluation performed at basal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prediabetes, defined for the existence impaired glucose tolerance (glucose between 140 and 199 mg/dL at the 2 hours of the Oral Tolerance Glucose Test (OGTT) with impaired fasting glucose (fasting glucose between 100 and 125 mg/dL)
* Patients who accept to participate in the study and sign the informed consent letter.

Exclusion Criteria:

* Patients with diagnosed Type 2 Diabetes previously or detected during the OGTT
* Patients in actual treatment or during the last 3 months with metformin, pioglitazone or another antidiabetic drug, including insulin
* Serum creatinine > 1.6 mg/dL
* Hypertriglyceridemia very high (>500 mg/dL)
* Pregnant women
* Altered arterial hypertension (Systolic >180 mmHg or Diastolic >105 mmHg)
* Excessive alcohol intake, acute or chronic
* Medications or medical conditions that affect glucose homeostasis (thiazides, beta blockers, glucocorticoids for systemic use, weight-reducing drugs or anorexigenics, Cushing´s syndrome, thyrotoxicosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from basal fasting and post2h OGTT glucose levels at 6 and 12 months | 6 and 12 months
  Fasting and post-2h OGTT glucose values (mg/dl)

SECONDARY OUTCOMES:
Change from basal pancreatic beta cell function at 6 and 12 months | 6 and 12 months
  Evaluated with the measurements of glucose and insulin during the oral glucose tolerance
Change from basal insulin sensitivity at 6 and 12 months | 6 and 12 months
  Insulin sensitivity evaluated during the oral glucose tolerance test by Matsuda index
Change from basal Weight at 6 and 12 months | 6 and 12 months
  Weight measurement during the study, in kg

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Guardado-Mendoza, MDPhD, Principal Investigator — Universidad de Guanajuato
Locations (1):
- Universidad de Guanajuato, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No
Data collection could be shared by the principal investigator on a particular request

REFERENCES:
- [Background] Juarez-Rojop IE, Fortuny-Falconi CM, Gonzalez-Castro TB, Tovilla-Zarate CA, Villar-Soto M, Sanchez ER, Hernandez-Diaz Y, Lopez-Narvaez ML, Ble-Castillo JL, Perez-Hernandez N, Rodriguez-Perez JM. Association between reduced quality of life and depression in patients with type 2 diabetes mellitus: a cohort study in a Mexican population. Neuropsychiatr Dis Treat. 2018 Oct 4;14:2511-2518. doi: 10.2147/NDT.S167622. eCollection 2018. PMID 30323600
- [Background] van Dieren S, Beulens JW, van der Schouw YT, Grobbee DE, Neal B. The global burden of diabetes and its complications: an emerging pandemic. Eur J Cardiovasc Prev Rehabil. 2010 May;17 Suppl 1:S3-8. doi: 10.1097/01.hjr.0000368191.86614.5a. PMID 20489418
- [Background] Lupi R, Del Prato S. Beta-cell apoptosis in type 2 diabetes: quantitative and functional consequences. Diabetes Metab. 2008 Feb;34 Suppl 2:S56-64. doi: 10.1016/S1262-3636(08)73396-2. PMID 18640587
- [Background] Huang Y, Cai X, Chen P, Mai W, Tang H, Huang Y, Hu Y. Associations of prediabetes with all-cause and cardiovascular mortality: a meta-analysis. Ann Med. 2014 Dec;46(8):684-92. doi: 10.3109/07853890.2014.955051. Epub 2014 Sep 18. PMID 25230915
- [Background] Sun ZJ, Yang YC, Wu JS, Wang MC, Chang CJ, Lu FH. Increased risk of glomerular hyperfiltration in subjects with impaired glucose tolerance and newly diagnosed diabetes. Nephrol Dial Transplant. 2016 Aug;31(8):1295-301. doi: 10.1093/ndt/gfv385. Epub 2015 Nov 25. PMID 26610595
- [Background] Butler AE, Janson J, Bonner-Weir S, Ritzel R, Rizza RA, Butler PC. Beta-cell deficit and increased beta-cell apoptosis in humans with type 2 diabetes. Diabetes. 2003 Jan;52(1):102-10. doi: 10.2337/diabetes.52.1.102. PMID 12502499
- [Background] Martin BC, Warram JH, Krolewski AS, Bergman RN, Soeldner JS, Kahn CR. Role of glucose and insulin resistance in development of type 2 diabetes mellitus: results of a 25-year follow-up study. Lancet. 1992 Oct 17;340(8825):925-9. doi: 10.1016/0140-6736(92)92814-v. PMID 1357346
- [Background] Ferrannini E. Insulin resistance versus beta-cell dysfunction in the pathogenesis of type 2 diabetes. Curr Diab Rep. 2009 Jun;9(3):188-9. doi: 10.1007/s11892-009-0031-8. No abstract available. PMID 19490819
- [Background] Gastaldelli A, Ferrannini E, Miyazaki Y, Matsuda M, DeFronzo RA; San Antonio metabolism study. Beta-cell dysfunction and glucose intolerance: results from the San Antonio metabolism (SAM) study. Diabetologia. 2004 Jan;47(1):31-9. doi: 10.1007/s00125-003-1263-9. Epub 2003 Dec 10. PMID 14666364
- [Background] Dunning BE, Gerich JE. The role of alpha-cell dysregulation in fasting and postprandial hyperglycemia in type 2 diabetes and therapeutic implications. Endocr Rev. 2007 May;28(3):253-83. doi: 10.1210/er.2006-0026. Epub 2007 Apr 4. PMID 17409288
- [Background] Nauck MA, El-Ouaghlidi A, Gabrys B, Hucking K, Holst JJ, Deacon CF, Gallwitz B, Schmidt WE, Meier JJ. Secretion of incretin hormones (GIP and GLP-1) and incretin effect after oral glucose in first-degree relatives of patients with type 2 diabetes. Regul Pept. 2004 Nov 15;122(3):209-17. doi: 10.1016/j.regpep.2004.06.020. PMID 15491793
- [Background] Enoki S, Mitsukawa T, Takemura J, Nakazato M, Aburaya J, Toshimori H, Matsukara S. Plasma islet amyloid polypeptide levels in obesity, impaired glucose tolerance and non-insulin-dependent diabetes mellitus. Diabetes Res Clin Pract. 1992 Jan;15(1):97-102. doi: 10.1016/0168-8227(92)90074-2. PMID 1541241
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S13-S28. doi: 10.2337/dc19-S002. PMID 30559228
- [Background] Ascaso JF, Romero P, Real JT, Priego A, Valdecabres C, Carmena R. [Insulin resistance quantification by fasting insulin plasma values and HOMA index in a non-diabetic population]. Med Clin (Barc). 2001 Nov 3;117(14):530-3. doi: 10.1016/s0025-7753(01)72168-9. Spanish. PMID 11707218
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Background] Pan XR, Li GW, Hu YH, Wang JX, Yang WY, An ZX, Hu ZX, Lin J, Xiao JZ, Cao HB, Liu PA, Jiang XG, Jiang YY, Wang JP, Zheng H, Zhang H, Bennett PH, Howard BV. Effects of diet and exercise in preventing NIDDM in people with impaired glucose tolerance. The Da Qing IGT and Diabetes Study. Diabetes Care. 1997 Apr;20(4):537-44. doi: 10.2337/diacare.20.4.537. PMID 9096977
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Defronzo RA, Banerji M, Bray GA, Buchanan TA, Clement S, Henry RR, Kitabchi AE, Mudaliar S, Musi N, Ratner R, Reaven PD, Schwenke D, Stentz FB, Tripathy D. Actos Now for the prevention of diabetes (ACT NOW) study. BMC Endocr Disord. 2009 Jul 29;9:17. doi: 10.1186/1472-6823-9-17. PMID 19640291
- [Background] Drucker DJ, Sherman SI, Gorelick FS, Bergenstal RM, Sherwin RS, Buse JB. Incretin-based therapies for the treatment of type 2 diabetes: evaluation of the risks and benefits. Diabetes Care. 2010 Feb;33(2):428-33. doi: 10.2337/dc09-1499. No abstract available. PMID 20103558
- [Background] Lundkvist P, Pereira MJ, Katsogiannos P, Sjostrom CD, Johnsson E, Eriksson JW. Dapagliflozin once daily plus exenatide once weekly in obese adults without diabetes: Sustained reductions in body weight, glycaemia and blood pressure over 1 year. Diabetes Obes Metab. 2017 Sep;19(9):1276-1288. doi: 10.1111/dom.12954. Epub 2017 May 31. PMID 28345814
- [Background] Abdul-Ghani M, Al Jobori H, Daniele G, Adams J, Cersosimo E, Triplitt C, DeFronzo RA. Inhibition of Renal Sodium-Glucose Cotransport With Empagliflozin Lowers Fasting Plasma Glucose and Improves beta-Cell Function in Subjects With Impaired Fasting Glucose. Diabetes. 2017 Sep;66(9):2495-2502. doi: 10.2337/db17-0055. Epub 2017 Jun 13. PMID 28611037
- [Background] Ferrannini E, Mark M, Mayoux E. CV Protection in the EMPA-REG OUTCOME Trial: A "Thrifty Substrate" Hypothesis. Diabetes Care. 2016 Jul;39(7):1108-14. doi: 10.2337/dc16-0330. PMID 27289126
- [Background] Packer M, Anker SD, Butler J, Filippatos G, Zannad F. Effects of Sodium-Glucose Cotransporter 2 Inhibitors for the Treatment of Patients With Heart Failure: Proposal of a Novel Mechanism of Action. JAMA Cardiol. 2017 Sep 1;2(9):1025-1029. doi: 10.1001/jamacardio.2017.2275. PMID 28768320
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Gonzalez-Heredia T, Hernandez-Corona DM, Gonzalez-Ortiz M, Martinez-Abundis E. Effect of Linagliptin Versus Metformin on Glycemic Variability in Patients with Impaired Glucose Tolerance. Diabetes Technol Ther. 2017 Aug;19(8):471-475. doi: 10.1089/dia.2017.0020. Epub 2017 Jun 5. PMID 28581818
- [Background] Lingvay I. SODIUM GLUCOSE COTRANSPORTER 2 AND DIPEPTIDYL PEPTIDASE-4 INHIBITION: PROMISE OF A DYNAMIC DUO. Endocr Pract. 2017 Jul;23(7):831-840. doi: 10.4158/EP161725.RA. Epub 2017 Mar 23. PMID 28332871

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT04131582/Prot_SAP_000.pdf